CLINICAL TRIAL: NCT01550250
Title: Feasibility of Night-time Compression Systems for Breast Cancer Related Lymphedema: a Pilot Study
Brief Title: Night-time Compression Systems for Breast Cancer Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other); Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACREC-25845
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Breast Neoplasms; Lymphedema
Keywords: Breast cancer; Arm lymphedema; Compression therapy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Night-time Compression (Experimental): Women randomized to the immediate night-time compression system group will be measured for a custom-made night-time compression system. Women in this group will be instructed to wear their night-time compression system garment for a minimum of 5 nights per week over the 12-week intervention period. A gradual increase in nights worn and wear-time of the garment will occur over the first two weeks. From weeks 3 to 12 of the study, the participants will be asked to wear the garment for 8 hours per night, for a minimum of five nights per week.
  Interventions: Behavioral: Night-time compression system garment; Behavioral: Day-time compression sleeve
- Delayed Group: Standard Care (Active Comparator): Women randomized to the delayed night-time compression system group will receive standard care for lymphedema maintenance. Each participant will be instructed to wear their day-time compression sleeve with or without a glove/ gauntlet, providing a minimum of 30 mm Hg of pressure, for twelve hours per day, each day of the week. Following the twelve-week delay period, women in this arm of the trial will be fitted for their respective night-time compression system garment and will follow the protocol outlined in the experimental arm of the trial.
  Interventions: Behavioral: Day-time compression sleeve

INTERVENTIONS:
Behavioral: Night-time compression system garment — Night-time compression system garment 8 hours per night for a minimum of 5 nights per week.
  Arms: Immediate Night-time Compression
Behavioral: Day-time compression sleeve — Standard care for lymphedema maintenance. Day-time compression sleeve with or without a glove/ gauntlet, providing a minimum of 30 mm Hg of pressure, for twelve hours per day, each day of the week.

SUMMARY:
Women who have undergone breast cancer surgery may develop swelling of the arm on the side the breast cancer occurred. If the swelling becomes chronic it is called lymphedema. This study will examine night-time compression system garments for lymphedema. Our objective is to determine if breast cancer survivors are willing and able to use the garment overnight to help control their lymphedema. Thirty breast cancer survivors from Alberta will be enrolled in the 24-week long study. Measurements will be taken of each arm to assess the extent of lymphedema and to measure changes over the study period. We will also examine other outcomes such as the impact of the night-time compression system garment on sleep. The study will provide important information on the feasibility of night-time compression system garments as a self-management strategy for lymphedema.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a histological diagnosis of breast cancer experiencing edema in the ipsilateral arm such that there is a minimum 10% and maximum 40% increase in arm volume over the unaffected arm (mild to moderate lymphedema).
2. Patients must have completed all primary and adjuvant treatments (surgery, chemotherapy, radiotherapy) prior to randomization.
3. Patients must have their own fitted compression garment for daytime maintenance.
4. No past or current use of a night-time compression system for maintenance. Those patients who have trialed a night-time compression system in the past year must observe a six-month washout period before entering the trial.

Exclusion Criteria:

1. Clinical or radiological evidence of active disease, either local or metastatic.
2. History of contralateral breast cancer and axillary surgery.
3. Serious non-malignant disease, such as renal or cardiac failure, which would preclude daily treatment and follow-up.
4. Patients for whom compression is contraindicated.
5. Psychiatric or addictive disorders which preclude obtaining informed consent or adherence to the protocol.
6. Unable to comply with the protocol, measurement and follow-up schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Accrual rate | 18 months
  The number of women eligible for the study and number agreeing to participate.

SECONDARY OUTCOMES:
Adherence | 24 weeks
  Data on adherence to wearing the night-time compression system.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L. McNeely, PhD, Principal Investigator — University of Alberta and Alberta Health Services
Locations (2):
- Canada (2):
  - Holy Cross Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta